CLINICAL TRIAL: NCT01622634
Title: The E-PHIT Study: Eggs, Protein, and High-Intensity Training: A Diabetes Prevention Program for Women
Brief Title: Effect of a High-Protein Diet and/or High-Intensity Training on Metabolic Syndrome
Acronym: EPHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Ellen Evans, Associate Professor, Principal Investigator, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPHIT
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Metabolic Syndrome
Keywords: cardiovascular disease; diabetes mellitus
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Higher Protein Diet (PRO) (Active Comparator)
  Interventions: Other: Higher PRO Diet
- Higher Carbohydrate Diet (CARB) (Active Comparator)
  Interventions: Other: Higher CARB Diet
- PRO & Interval Exercise (PRO+EX) (Active Comparator)
  Interventions: Behavioral: Sprint Interval Exercise; Other: Higher PRO Diet
- CARB & Interval Exercise (CARB+EX) (Active Comparator)
  Interventions: Behavioral: Sprint Interval Exercise; Other: Higher CARB Diet

INTERVENTIONS:
Behavioral: Sprint Interval Exercise — Participants will undergo sprint interval training on a cycle ergometer 3 times weekly for 6 weeks. Each training session begins with a 5-minute active warm-up. The warm-up is followed by 4-7 bouts of 30 seconds of all-out sprints and 4 minutes of active recovery.
  Other Names: High Intensity Training; Sprint Interval Cycling
  Arms: CARB & Interval Exercise (CARB+EX); PRO & Interval Exercise (PRO+EX)
Other: Higher PRO Diet — Participants in the PRO and PRO+EX groups will meet weekly with a diet specialist on staff to monitor their intake and compliance with the high protein diet.
  Other Names: Higher Protein Reduced Carbohydrate Diet
  Arms: Higher Protein Diet (PRO); PRO & Interval Exercise (PRO+EX)
Other: Higher CARB Diet — Participants in the CHO and CHO+EX groups will meet weekly with a diet specialist on staff to monitor their intake and compliance with the higher carbohydrate diet.
  Other Names: Conventional Higher Carbohydrate Diet
  Arms: CARB & Interval Exercise (CARB+EX); Higher Carbohydrate Diet (CARB)

SUMMARY:
The objective of this study is to determine the combined effects of a high-protein diet and high-intensity training on metabolic syndrome risk factors in women aged 30-65.

DETAILED DESCRIPTION:
High-protein diet interventions have been shown to be effective in reducing triglycerides and increasing high-density lipoprotein cholesterol concentrations. Low-volume, high-intensity cycling exercise has shown to elicit positive effects on metabolic syndrome risk factors such as triglyceride concentrations. The objective of this study was to determine the combined effects of a high-protein, reduced carbohydrate diet and high-intensity interval training on metabolic syndrome risk factors in women. The second primary aim is to investigate the effect of the macronutrient content of the post-exercise meal consumed following an acute bout of interval training on postprandial metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-65 yrs of age, inclusive
* Waist circumference > 88 cm.
* Weight stable (within 2 kg) for past 6 mo
* Sedentary/Low-active (defined as <300minutes/wk light or moderate activity, with no vigorous activity in last 6 months)
* At risk for MetS [defined as having 2 of the following 4 factors: 1) hypertriglyceridemia defined as > 150 mg/mL, 2) low HDL cholesterol defined < 50 or on medication, 3) elevated blood pressure defined as > 130/>85 Hg or taking medications or 4) hyperglycemia defined as fasting blood glucose > 100 or glycated hemoglobin > 6.5 or taking medications.
* Willing to be randomized to the four treatment groups

Exclusion Criteria:

* Any chronic disease/condition that would not permit exercise or dietary restriction (including egg allergy or refusal to incorporate eggs into the diet) or alter interpretation of data. Examples include, but are not limited to:

  1. cardiopulmonary disease (e.g. recent myocardial infarction, unstable angina, stroke) or unstable disease; 2) severe orthopedic, musculoskeletal or neuromuscular impairments that would contradict exercise; 3) sensory impairments that interfere with following directions; 4) diagnosis of dementia; 5) history of malignancy during the past 5 yr; 6) medication use that impacts primary outcomes of interest (e.g. statins); 7) weight greater than 400 pounds due to DXA weight and size limitations; 8) Uncontrolled blood pressure defined as > 160/>100 Hg.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome Risk Factors | Change [Baseline to 6 Weeks]
  1. Post-Prandial Lipemia (and/or metabolic responses including insulin, glucose, triglycerides and free-fatty acids) to: a) a high fat meal challenge and b) a meal challenge similar to the higher protein or carbohydrate treatment arm. After an overnight fast and baseline blood draws, participants will consume a small meal and have their blood sampled every 30 minutes for 3 hours.
  2. Biomarkers for Cardiovascular Disease and Diabetes Mellitus. Fasting blood samples for serum lipids, glucose, insulin and systemic inflammation (C-reactive protein) will be taken after an overnight fast.

SECONDARY OUTCOMES:
Satiety | Change [Baseline to 6 weeks]
  Satiety will be assessed using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M. Evans, PhD, Principal Investigator — University of Georgia; Kirk J. Cureton, PhD, Principal Investigator — University of Georgia
Locations (1):
- Body Composition and Metabolism Lab, Ramsey Center, University of Georgia, Athens, Georgia, United States